CLINICAL TRIAL: NCT00002896
Title: RANDOMIZED TRIAL OF CONCOMITANT PREOPERATIVE RADIO-CHEMOTHERAPY WITH OR WITHOUT POSTOPERATIVE CHEMOTHERAPY IN LOCALLY ADVANCED RECTAL CARCINOMA
Brief Title: Radiation Therapy Plus Chemotherapy Before Surgery With or Without Chemotherapy After Surgery in Treating Patients With Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065222; CNR-9604; EU-96047
Record Dates: First submitted 1999-11-01; First posted 2004-05-13 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2008-02

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; recurrent rectal cancer; adenocarcinoma of the rectum; mucinous adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Drug Therapy; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: chemotherapy
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: conventional surgery
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, giving the drugs in different ways, and combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus fluorouracil and leucovorin before surgery given with or without fluorouracil and leucovorin after surgery in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the local recurrence rate, cost-benefit ratio, and acute and late toxicity associated with concomitant preoperative radiotherapy and fluorouracil/leucovorin (5-FU/CF) in patients with locally advanced adenocarcinoma of the rectum. II. Compare the relapse rate, survival rate, disease-free interval, and cost-benefit ratio associated with 6 courses of postoperative 5-FU/CF vs. no further treatment in these patients.

OUTLINE: This is a randomized study. Patients are stratified by tumor stage, age, type of surgery, and participating institution. Patients are randomly assigned to one of two groups. The first group receives radiotherapy to the tumor over 5 weeks and concomitant fluorouracil/leucovorin for 5 consecutive days on the first and fifth weeks. Four to six weeks later, patients undergo complete resection, followed upon recovery by fluorouracil/leucovorin every 4 weeks for 6 courses. The second group receives preoperative chemoradiotherapy followed by surgery, as above, with no postoperative treatment. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 774 patients will be entered on this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma or mucinous adenocarcinoma of the rectum Distal limit of tumor no higher than 12 cm from the anal verge on proctoscopy Locally advanced (T3-4 M0) tumor by one of the following: Partial fixation Complete stenosis Invasion beyond the muscular stratum on transrectal ultrasound

PATIENT CHARACTERISTICS: Age: 75 and under Performance status: WHO 0 or 1 Hematopoietic: WBC greater than 3,000 Platelets greater than 130,000 Hepatic: Not specified Renal: Creatinine less than 1.4 mg/dL Cardiovascular: No unstable angina No cardiac decompensation Other: No prior or concurrent malignancy

PRIOR CONCURRENT THERAPY: Not specified

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 774 (Estimated)
Dates: Start 1993-09

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cionini, MD, Study Chair — Santa Chiara Hospital
Locations (1):
- Ospedale St. Santa Chiara, Pisa, Italy

REFERENCES:
- [Result] Cionini L, Cartei F, Manfredi B, et al.: Randomized study of preoperative chemoradiation (CTRT) in locally advanced rectal cancer: preliminary results. [Abstract] Int J Radiat Oncol Biol Phys 45 (3 Suppl): A-61, 178, 1999.